CLINICAL TRIAL: NCT05341596
Title: Incidence and Outcome of Reintubation in the Postanesthesia Care Unit: a Single-center, Retrospective, Observational Matched Cohort Study in China
Brief Title: Incidence and Outcome of Reintubation in the PACU
Status: Completed | Type: Observational
Sponsor: Shangkun Liu (200966) (Other)
Responsible Party: Sponsor-Investigator, Shangkun Liu (200966), nurse manager, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20170501
Record Dates: First submitted 2022-04-08; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Complications; Complication of Medical Care
Keywords: general anesthesia; postanesthesia care unit; reintubation after planned extubation
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reintubation after planned extubation: Reintubation after planned extubation(RAP) was defined as repeat endotracheal intubation in the PACU after planned extubation of the initial endotracheal intubation for general anesthesia or combined general anesthesia other than that performed in the operating room.
  Interventions: Procedure: repeat endotracheal intubation
- matched group: Patients without RAP during the PACU stay were designated as the matched group

INTERVENTIONS:
Procedure: repeat endotracheal intubation — repeat endotracheal intubation in the PACU after planned extubation of the initial endotracheal intubation for general anesthesia or combined general anesthesia other than that performed in the operating room
  Groups: Reintubation after planned extubation

SUMMARY:
This study evaluated the occurrence of reintubation after planned extubation (RAP), the impact of RAP on duration of PACU stay,length of stay,length of postoperative stay,inpatient healthcare costs, unanticipated ICU admission and readmission.

DETAILED DESCRIPTION:
The study was carried out in Wuhan City, China at a general public university hospital with 62 clinical departments, 99 surgical rooms, and 38 beds in the PACU. The total number of operations performed in this hospital is more than 90,000/year. The study was approved by the hospital ethics committee and was deemed that written patient consent was not required. The adverse events, including RAP, in all patients in the PACU were recorded on a standardized form in a database by pre-trained qualified nurses and/or anesthesiologists at the time of care from January 1, 2017 to December 31, 2019.

Data, including patient demographic and surgical and anesthesia parameters, were obtained from the anesthesia information system. Adverse events management and duration of PACU stay were also documented. For three years, all collected data were filed in a computer every day and were summarized and analyzed every month. Data, such as demographics, airway, oxygen saturation, consciousness, treatment, vital signs, and fast-track criteria scores, were recorded for all patients in the PACU. The first part contained preoperative and intraoperative data, which were entered into the database by the anesthesiologists involved in the patients' intraoperative care from the time of PACU admission. The second part were recorded by nurse and comprised postoperative data from the PACU to the ward or ICU. The third part were recorded by the surgeons and/ or surgical nurses and comprised postoperative data. The criteria for tracheal extubation in the operating room(OR) and the timing of transfer to the PACU were the responsibility of the anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring stay in PACU

Exclusion Criteria:

* Patients were transferred directly from the operating room to the ward or icu
* non-postoperative patient

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Reintubation after planned extubation was defined as repeat endotracheal intubation in the PACU after planned extubation of the initial endotracheal intubation for general anesthesia or combined general anesthesia other than that performed in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 121965 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Duration of PACU stay | through study completion, an average of three months
  From patient transfer into PACU to transfer out of PACU
Length of postoperative stay | through study completion, an average of three months
Unanticipated ICU admission | through study completion, an average of three months
  Unplanned transfer to the ICU

SECONDARY OUTCOMES:
Inpatient healthcare costs | through study completion, an average of three months
  Any medical cost during hospital stay
Length of stay | through study completion, an average of three months
  The time of hospital length of stay
Duration of postoperative monitoring | through study completion, an average of three months
  The time of postoperative monitoring
Readmission | through study completion, an average of three months
  admission after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hui Xu, Study Chair — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No
Reintubation after planned extubation (RAP) is a serious adverse event. This study aimed to determine the rate and impact of RAP on postoperative course and hospitalization outcomes

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Postanesthetic Care. Practice guidelines for postanesthetic care: a report by the American Society of Anesthesiologists Task Force on Postanesthetic Care. Anesthesiology. 2002 Mar;96(3):742-52. doi: 10.1097/00000542-200203000-00033. No abstract available. PMID 11873052
- [Background] Tarrac SE. A description of intraoperative and postanesthesia complication rates. J Perianesth Nurs. 2006 Apr;21(2):88-96. doi: 10.1016/j.jopan.2006.01.006. PMID 16600829
- [Background] Siddiqui N, Arzola C, Teresi J, Fox G, Guerina L, Friedman Z. Predictors of desaturation in the postoperative anesthesia care unit: an observational study. J Clin Anesth. 2013 Dec;25(8):612-7. doi: 10.1016/j.jclinane.2013.04.018. Epub 2013 Oct 4. PMID 24095886
- [Background] Rujirojindakul P, Geater AF, McNeil EB, Vasinanukorn P, Prathep S, Asim W, Naklongdee J. Risk factors for reintubation in the post-anaesthetic care unit: a case-control study. Br J Anaesth. 2012 Oct;109(4):636-42. doi: 10.1093/bja/aes226. Epub 2012 Jul 9. PMID 22777658
- [Background] Haritos G, Smith CA, Haas RE, Becker A, Nguyen D, Stierer KA, Klein M. Critical Events Leading to Endotracheal Reintubation in the Postanesthesia Care Unit: A Retrospective Inquiry of Contributory Factors. AANA J. 2019 Feb;87(1):59-63. PMID 31587745
- [Background] Lee PJ, MacLennan A, Naughton NN, O'Reilly M. An analysis of reintubations from a quality assurance database of 152,000 cases. J Clin Anesth. 2003 Dec;15(8):575-81. doi: 10.1016/j.jclinane.2003.03.006. PMID 14724078
- [Background] Bruins SD, Leong PM, Ng SY. Retrospective review of critical incidents in the post-anaesthesia care unit at a major tertiary hospital. Singapore Med J. 2017 Aug;58(8):497-501. doi: 10.11622/smedj.2016126. Epub 2016 Jul 21. PMID 27439784
- [Background] Ting PC, Chou AH, Yang MW, Ho AC, Chang CJ, Chang SC. Postoperative reintubation after planned extubation: a review of 137,866 general anesthetics from 2005 to 2007 in a Medical Center of Taiwan. Acta Anaesthesiol Taiwan. 2010 Dec;48(4):167-71. doi: 10.1016/j.aat.2010.12.003. Epub 2010 Dec 22. PMID 21195986
- [Background] Siao-feng A, Tai-di Z, OU QH. Risk factors for postoperative reintubation in patients undergoing general anesthesia. Chin J Anesthesiol. 2013;33(12):1427-30.
- [Background] Beverly A, Brovman EY, Malapero RJ, Lekowski RW, Urman RD. Unplanned Reintubation Following Cardiac Surgery: Incidence, Timing, Risk Factors, and Outcomes. J Cardiothorac Vasc Anesth. 2016 Dec;30(6):1523-1529. doi: 10.1053/j.jvca.2016.05.033. Epub 2016 May 21. PMID 27595531
- [Background] Menon N, Joffe AM, Deem S, Yanez ND, Grabinsky A, Dagal AH, Daniel S, Treggiari MM. Occurrence and complications of tracheal reintubation in critically ill adults. Respir Care. 2012 Oct;57(10):1555-63. doi: 10.4187/respcare.01617. Epub 2012 Feb 10. PMID 22324979
- [Background] Ing C, Chui I, Ohkawa S, Kakavouli A, Sun L. Incidence and causes of perioperative endotracheal reintubation in children: a review of 28,208 anesthetics. Paediatr Anaesth. 2013 Jul;23(7):621-6. doi: 10.1111/j.1460-9592.2012.03920.x. Epub 2012 Jul 23. PMID 22817271
- [Background] De la Garza Ramos R, Passias PG, Schwab F, Bydon A, Lafage V, Sciubba DM. Incidence, Risk Factors, and Mortality of Reintubation in Adult Spinal Deformity Surgery. Clin Spine Surg. 2017 Aug;30(7):E896-E900. doi: 10.1097/BSD.0000000000000404. PMID 27352366
- [Background] Gao F, Yang LH, He HR, Ma XC, Lu J, Zhai YJ, Guo LT, Wang X, Zheng J. The effect of reintubation on ventilator-associated pneumonia and mortality among mechanically ventilated patients with intubation: A systematic review and meta-analysis. Heart Lung. 2016 Jul-Aug;45(4):363-71. doi: 10.1016/j.hrtlng.2016.04.006. PMID 27377334
- [Result] Liu SK, Chen G, Yan B, Huang J, Xu H. Adverse Respiratory Events Increase Post-anesthesia Care Unit Stay in China: A 2-year Retrospective Matched Cohort Study. Curr Med Sci. 2019 Apr;39(2):325-329. doi: 10.1007/s11596-019-2038-y. Epub 2019 Apr 23. PMID 31016529